CLINICAL TRIAL: NCT02117024
Title: A Phase 2, Multicenter, Randomized Study to Evaluate the Safety and Efficacy of Viagenpumatucel-L (HS-110) in Combination With Low Dose (Metronomic) Cyclophosphamide Versus Chemotherapy Alone in Patients With Non-Small Cell Lung Adenocarcinoma After Failure of Two or Three Previous Treatment Regimens for Advanced Disease
Brief Title: A Phase 2 Study of Viagenpumatucel-L (HS-110) in Patients With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision; strategic - based on changing treatment landscape
Sponsor: Heat Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS110-201
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung; cancer; gp96; vaccine; immunotherapy; Heat Biologics; cyclophosphamide; vinorelbine; erlotinib; gemcitabine; paclitaxel; docetaxel; pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Vinorelbine; Erlotinib Hydrochloride; Gemcitabine; Paclitaxel; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viagenpumatucel-L Plus Metronomic Cyclophosphamide (Experimental): Viagenpumatucel-L (HS-110) given as 1*10^7 cells for 12 weekly injections followed by injections every 9 weeks for up to 12 months or until discontinuation from study treatment, whichever occurs first, plus metronomic cyclophosphamide therapy for the first 12 weeks.
  Interventions: Drug: Viagenpumatucel-L; Drug: Metronomic Cyclophosphamide
- Chemotherapy Alone (Active Comparator): Patients will be treated with a physician's choice regimen until progression.
  Interventions: Drug: Physician's Choice Regimen (Vinorelbine, Erlotinib, Gemcitabine, Paclitaxel, Docetaxel, Pemetrexed)

INTERVENTIONS:
Drug: Viagenpumatucel-L — Vaccine derived from irradiated human lung cancer cells genetically engineered to continually secrete gp96-Ig
  Other Names: HS-110
  Arms: Viagenpumatucel-L Plus Metronomic Cyclophosphamide
Drug: Metronomic Cyclophosphamide — One 50mg tablet administered orally daily for 7 days on alternating weeks for a total of 6 weeks of therapy over 12 weeks
  Arms: Viagenpumatucel-L Plus Metronomic Cyclophosphamide
Drug: Physician's Choice Regimen (Vinorelbine, Erlotinib, Gemcitabine, Paclitaxel, Docetaxel, Pemetrexed) — Physician will select one of the following to be given in nominal 21 day cycles with dose and route according to investigator's standard practice:
  * Vinorelbine
  * Erlotinib
  * Gemcitabine
  * Paclitaxel
  * Docetaxel
  * Pemetrexed
  Arms: Chemotherapy Alone

SUMMARY:
Determine whether viagenpumatucel-L combined with low-dose cyclophosphamide prolongs survival in patients with NSCLC who failed 2 or 3 prior lines of therapy for incurable or metastatic disease compared with chemotherapy alone.

DETAILED DESCRIPTION:
This study will test whether vaccination with viagenpumatucel-L combined with low-dose cyclophosphamide will prolong the survival of patients with non-small cell lung cancer (NSCLC) who have failed 2 or 3 prior lines of therapy for incurable or metastatic disease compared with chemotherapy alone. Patients will be randomized 2 to 1 into the viagenpumatucel-L arm and the chemotherapy alone arm, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung adenocarcinoma
* At least 2 and no more than 3 prior lines of therapy for incurable or metastatic NSCLC
* Suitable for conventional single agent chemotherapy
* Disease progression at study entry
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1; PS=2 patients may be considered
* Central nervous system (CNS) metastases may be permitted but must be treated and neurologically stable
* Adequate laboratory parameters
* Willing and able to comply with the protocol and sign informed consent
* Female patients who are of childbearing potential and fertile male patients must agree to use an effective form of contraception throughout study participation

Exclusion Criteria:

* Received systemic anticancer therapy or radiation therapy within the previous 14 days
* Received more than 3 lines of prior conventional therapy for advanced disease
* Human immunodeficiency virus (HIV), hepatitis B or C, or severe/uncontrolled infections or intercurrent illness, unrelated to the tumor, requiring active therapy
* Any condition requiring concurrent systemic immunosuppressive therapy
* Known immunodeficiency disorders
* Known leptomeningeal disease
* Other active malignancies
* Prior treatment with a cancer vaccine for this indication
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-07; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Cohen, MD, Principal Investigator — University of Pennsylvania
Locations (16):
- United States (16):
  - Highlands Oncology Group, Rogers, Arkansas
  - University of California San Diego, La Jolla, California
  - University of California at Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - Georgia Regents University, Augusta, Georgia
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Syracuse, Syracuse, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Providence Portland Medical Center- Providence Lung Cancer Clinic, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Oncology PA Texas Cancer Center, Abilene, Texas
  - Mary Crowley Cancer Center, Dallas, Texas
  - Cancer Care Northwest, Spokane, Washington
  - Aurora Research Institute, Green Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy Alone: Patients will be treated with a physician's choice regimen until progression.
  Physician's Choice Regimen (Vinorelbine, Erlotinib, Gemcitabine, Paclitaxel, Docetaxel, Pemetrexed): Physician will select one of the following to be given in nominal 21 day cycles with dose and route according to investigator's standard practice:
  * Vinorelbine
  * Erlotinib
  * Gemcitabine
  * Paclitaxel
  * Docetaxel
  * Pemetrexed
Period: Overall Study
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Started | 45 | 21
Completed | 1 | 1
Not Completed | 44 | 20
Not completed — Progressive Disease | 26 | 9
Not completed — Significant Clinical Progression | 7 | 4
Not completed — Death | 5 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Randomized in Error | 1 | 0
Not completed — Patient returned to primary oncologist | 0 | 1
Not completed — Patient took treatment break | 0 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: Sixty-six of the original 123 planned patients were enrolled from June 2014 to 10 September 2015. Patients were randomized in a 2:1 ratio in the experimental group (n=45) and the control group (n=21). Sixty-three patients were included in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone | Total
Number analyzed (Participants) | 45 | 21 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 12 | 33
  >=65 years | 24 | 9 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.9) | 63.0 (10.5) | 64.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 10 | 37
  Male | 18 | 11 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 44 | 21 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 44 | 18 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 18 | 56
  Australia | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) calculated as the duration of survival from the date of randomization to the date of death from any cause, or was censored on the date the patient was last known to be alive.
  Survival time was calculated from the randomization date up to the date of death,or censored on the date that the patient was last known to be alive (last available visit date) utilizing Kaplan-Meier Estimate of Overall Survival Ending Events
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 45 | 21
Days | 176 [114.0 to 231.0] | 372 [204.0 to 875.0]
Statistical Analysis 1: Comparison: Viagenpumatucel-L Plus Metronomic Cyclophosphamide vs Chemotherapy Alone; Test type: Superiority; p = 0.0011, Log Rank
Statistical Analysis 2: Comparison: Viagenpumatucel-L Plus Metronomic Cyclophosphamide vs Chemotherapy Alone; With only 50% of enrollment complete prior to study termination by sponsor, insufficient sample size exists to fully complete efficacy analysis; Test type: Other; p < 0.05, Other; Hazard Ratio (HR) = 1.0

2. Secondary Outcome: Frequency of Adverse Events: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: Evaluate the safety of the combination of viagenpumatucel-L and low-dose cyclophosphamide by frequency of Treatment-Emergent Adverse Events
Time Frame: Up to 3 years
Population: Safety was defined as the number of adverse events (AE)/serious adverse events (SAE) in patients receiving viagenpumatucel-L and low-dose Cyclophosphamide (CY).
Measure: Count of Participants; unit: Participants
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 43 | 20
Participants
  At least one TEAE | 41 | 20
  At least one severe TEAE | 25 | 11
  At least one treatment-related TEAE | 32 | 15
  At least one SAE | 17 | 8
  Fatal TEAE | 7 | 0
  At least one TEAE Leading to Tx Discontinuation | 7 | 2
  At least one TEAE Leading to a Dose Reduction | 0 | 2

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Evaluate overall immune-related DCR (irDCR) and also DCR by Response Evaluation Criteria in Solid Tumors (RECIST) (complete response, partial response, and stable disease)
Time Frame: Up to 3 years
Population: Data were not collected for Outcome Measure 3 due to study termination (50% enrollment) by the Sponsor on 01 September 2015 due to changing treatment landscape (PD-1 approvals), and a subsequent change in development focus to Immuno-Oncology (IO) combinations. See NCT02439450.
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: 6-Month Disease Control Rate (6mDCR)
Description: Evaluate 6-month immune-related DCR (6m-irDCR) and also 6mDCR by RECIST (complete response, partial response, and stable disease at 6 months following randomization)
Time Frame: 6 months
Population: Data were not collected for Outcome Measure 4 due to study termination (50% enrollment) by the Sponsor on 01 September 2015 due to changing treatment landscape (PD-1 approvals), and a subsequent change in development focus to Immuno-Oncology (IO) combinations. See NCT02439450.
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Response Rate (ORR)
Description: Evaluate immune-related ORR (irORR) and also ORR by RECIST (complete response and partial response)
Time Frame: Up to 3 years
Population: Data were not collected for Outcome Measure 5 due to study termination (50% enrollment) by the Sponsor on 01 September 2015 due to changing treatment landscape (PD-1 approvals), and a subsequent change in development focus to Immuno-Oncology (IO) combinations. See NCT02439450.
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: Evaluate immune-related PFS (irPFS) and PFS by RECIST (Response Evaluation Criteria for Solid Tumors)
Time Frame: Up to 3 years
Population: Calculated from randomization date to earliest date of first 'Progressive Disease' response (Immune-Related / RECIST Response Criteria) or date of death, and censored on the date of the last available post-baseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 45 | 21
Days
  immune-related PFS (irPFS) | 76.0 [66.0 to 106.0] | 190.0 [72.0 to 445.0]
  Progression Free Survival (PFS) | 70.0 [65.0 to 96.0] | 190.0 [72.0 to 317.0]

7. Secondary Outcome: Time to Progression (TTP)
Description: Evaluate immune-related TTP (irTTP) and also TTP (Time to Progression) by RECIST
Time Frame: Up to 3 years
Population: Time to immune-related progression was calculated from the randomization date up to the date of the first 'Progressive Disease' response (Immune-Related Response Criteria) Time to progression was calculated from the randomization date up to the date of the first 'Progressive Disease' response (RECIST Response Criteria).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 45 | 21
Days
  immune-related TTP (irTTP) | 67.0 [61.0 to 76.0] | 71.0 [64.0 to 155.0]
  Time to Progression (TTP) | 67.5 [64.0 to 76.0] | 73.5 [64.0 to 198.0]

8. Secondary Outcome: Survival at 6 Months
Description: Evaluate the proportion of patients who are alive at 6 months following randomization
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 45 | 21
Participants | 21 | 17

9. Secondary Outcome: Survival at 12 Months
Description: Evaluate the proportion of patients who are alive at 12 months following randomization
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 45 | 21
Participants | 8 | 11

10. Secondary Outcome: Immune Response
Description: Characterize the peripheral blood immunologic response via intracellular cytokine staining (ICS) by flow cytometry and/or enzyme-linked immunosorbent spot (ELISPOT) on cluster of differentiation 8 positive (CD8+) cells following vaccination
Time Frame: Up to 3 years
Population: Data were not collected for Outcome Measure 10 due to study termination (50% enrollment) by the Sponsor on 01 September 2015 due to changing treatment landscape (PD-1 approvals), and a subsequent change in development focus to Immuno-Oncology (IO) combinations. See NCT02439450.
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year and 5 months
Arm/Group | Viagenpumatucel-L Plus Metronomic Cyclophosphamide | Chemotherapy Alone
All-Cause Mortality (participants affected / at risk) | 7/43 | 0/20
Serious Adverse Events (participants affected / at risk) | 17/43 | 8/20
Other Adverse Events (participants affected / at risk) | 19/43 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viagenpumatucel-L Plus Metronomic Cyclophosphamide (N=43) | Chemotherapy Alone (N=20)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Disease Progression (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Superior Vena Cava Syndrome (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viagenpumatucel-L Plus Metronomic Cyclophosphamide (N=43) | Chemotherapy Alone (N=20)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 7 (8)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Deep Vein Thrombosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hot Flush (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Superior Vena Cava Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was discontinued prematurely (50% enrollment) by the Sponsor on 01 September 2015 due to changing treatment landscape (PD-1 approvals), and a subsequent change in development focus to IO combinations. See NCT02439450.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT02117024/Prot_SAP_000.pdf